CLINICAL TRIAL: NCT06441968
Title: A Phase 1 Open-Label Safety and Immunogenicity Trial of MPV/S-2P, a Next Generation SARS-CoV-2 Booster Vaccine, in Previously Vaccinated Adults
Brief Title: Safety and Immunogenicity Trial of MPV/S-2P SARS-CoV-2 Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 23-1101
Record Dates: First submitted 2024-05-31; First posted 2024-06-04 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: adults; MPV/S-2P; phase 1; SARS-CoV-2; trial; vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Healthy adults between 18 - 64 years who have received a primary series and at least one booster with an authorized or licensed mRNA SARS-CoV-2 parenteral vaccine will receive 1 x 10^4 PFU of MPV/S-2P administered intranasally (approximately 0.5 mL per nostril) using VaxINator (Teleflex) for 1 year. N=20
  Interventions: Biological: MPV/S-2P
- Cohort 2 (Experimental): Healthy adults between 18 - 64 years who have received a primary series and at least one booster with an authorized or licensed mRNA SARS-CoV-2 parenteral vaccine will receive 1 x 10^5 PFU of MPV/S-2P administered intranasally (approximately 0.5 mL per nostril) using VaxINator (Teleflex) for 1 year. N=20
  Interventions: Biological: MPV/S-2P
- Cohort 3 (Experimental): Healthy adults between 18 - 64 years who have received a primary series and at least one booster with an authorized or licensed mRNA SARS-CoV-2 parenteral vaccine will receive 1 x 10^6 PFU of MPV/S-2P administered intranasally (approximately 0.5 mL per nostril) using VaxINator (Teleflex) for 1 year. N=20
  Interventions: Biological: MPV/S-2P

INTERVENTIONS:
Biological: MPV/S-2P — A live murine pneumonia virus (MPV) vector expressing an additional SARS-CoV-2 S-protein, stabilized in its prefusion form, is being tested for its efficacy in protecting against the SARS-CoV-2 virus. It is speculated to be a next-generation vaccine for COVID-19.

SUMMARY:
A clinical trial to evaluate the safety, reactogenicity, and immunogenicity of MPV/S-2P administered intranasally to adults who have previously received a primary series and at least one booster with an authorized or licensed mRNA SARS-CoV-2 parenteral vaccine. The primary objective is to evaluate the safety and reactogenicity of a single dose of MPV/S-2P in previously vaccinated healthy adults.

DETAILED DESCRIPTION:
A phase I clinical trial to evaluate the safety, reactogenicity, and immunogenicity of MPV/S-2P administered intranasally to adults who have previously received a primary series and at least one booster with an authorized or licensed mRNA SARS-CoV-2 parenteral vaccine. The study is designed as a non-randomized, open-label, dose-escalation clinical trial in non-pregnant adult participants, 18-64 years of age (with a goal of 30 percent or more >/=50 years of age), with or without prior SARS-CoV-2 infection, who are in good health and meet all other eligibility criteria. For the evaluation of three doses of MPV/S-2P vaccine, a sample size of 60 participants is anticipated.

To evaluate for early safety signals vaccination will proceed in a staged fashion. For Cohort 1, three sentinel participants under 50 years of age will be enrolled over at least 2 days. A safety review of clinical data and virologic shedding data through at least Day 8 will be conducted by the Safety Review Committee (SRC) prior to enrollment of the remainder of the cohort. Once Cohort 1 is fully enrolled, progression to Cohort 2 will be based on evaluation of halting rules, and cumulative clinical safety and virologic shedding data from Cohort 1 through at least Day 8 by the SRC.

Cohort 2 and 3 enrollment and safety oversight will proceed in the same fashion as Cohort 1. At the discretion of the SRC, additional participants in the cohort may be designated sentinels for any cohort. If halting rules are met the study will be paused for the SRC safety data review.

The primary objective is to evaluate the safety and reactogenicity of a single dose of MPV/S-2P in previously vaccinated healthy adults. The secondary objectives are 1) To evaluate the systemic anti-Spike humoral immune responses after vaccination 2) To evaluate nasal mucosal IgA and IgG responses after vaccination 3) To assess the duration and magnitude of viral vector (vaccine) shedding 4) To assess the immune response towards the vector.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to initiation of any study procedures.
2. Able to understand and agrees to comply with planned study procedures and be available for all study visits.
3. Non-pregnant adults, 18-64 years of age at time of vaccination.
4. Participants of childbearing potential * must agree to use or have practiced true abstinence ** or use at least one acceptable primary form of contraception *** * These criteria are applicable to persons assigned female at birth who have sexual intercourse with a person assigned male at birth, and who are of childbearing potential. Not of childbearing potential include post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure (R) placement) ** True abstinence is 100 percent of time no sexual intercourse (penis enters the vagina). Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods.

   *** Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the participant's vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable/transdermal hormonal birth control products. Must have used at least one acceptable primary form of contraception for at least 30 days prior to vaccination and agree to continue at least one acceptable primary form of contraception through 60 days after vaccination
5. Participants of childbearing potential must have a negative urine pregnancy test at screening and within 24 hours prior to study vaccination.
6. In general good health*.

   *As determined by medical history and physical examination, including vital signs, to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of safety of participants. Chronic medical diagnoses/ conditions should be stable for the last 30 days (i.e., no hospitalizations, ER, or urgent care for condition). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis/condition in the 30 days before study vaccination. Any prescription change that is due to change of health care provider, insurance company, etc., or done for financial reasons, and in the same class of medication, will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity.
7. Receipt of a complete primary COVID-19 mRNA vaccine series and at least one mRNA booster* with last vaccination at least 16 weeks prior to study vaccination.

   * Booster may be either homologous or heterologous to the primary vaccine series and must be an FDA authorized/licensed mRNA vaccine though doses may have been received as part of a clinical trial.
8. Clinical screening laboratory evaluations are within normal reference ranges or grade 1 with no clinical significance (NCS) per investigator discretion*.

   *White Blood Cells [WBCs] with differential, hemoglobin [Hgb], platelets [PLTs], Alanine Transaminase [ALT], Aspartate Transaminase [AST], Creatinine [Cr], Alkaline Phosphatase [ALP], Total Bilirubin [T. Bili]). ALT, AST, ALP, T. Bili and creatinine values that are below the reference range will not be exclusionary as these values below reference range are clinically insignificant.
9. Must agree to have samples stored for secondary research.
10. Must agree to wearing a surgical mask (or KN-95 or N-95) within 6 feet of others for 14 days after study vaccination, and potentially longer if asked by study team based on data gathered.

Exclusion Criteria:

1. Positive SARS-CoV-2 PCR at screening.
2. Abnormal vital signs (Grade 1 or higher)*

   *Grade 1 or higher is equivalent to: Systolic blood pressure (SBP) >/= 141 mmHg or </= 89 mmHg Diastolic blood pressure (DBP) >/= 91 mmHg Heart rate (HR) is >/= 101 beats per minute or </= 54 beats per minute Oral temperature >/= 38.0°C (100.4°F)
3. History of SARS-CoV-2 infection or receipt of any COVID-19 vaccine < 16 weeks prior to study vaccination.
4. Participant who is pregnant or breastfeeding.
5. Blood or plasma donation within 4 weeks prior to study vaccination.
6. Receipt of antibody or blood-derived products within 90 days prior to study vaccination.
7. Any self-reported or documented significant medical or psychiatric diseases* or any other condition that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation.

   *Significant medical or psychiatric conditions include but are not limited to respiratory disease (e.g., chronic obstructive pulmonary disease [COPD]) requiring daily medications currently, history of asthma in the past 5 years, or any treatment of respiratory disease exacerbations in the last 5 years. Significant kidney disease, liver disease, or cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), including any history of myocarditis or pericarditis, or uncontrolled cardiac arrhythmia. Neurological or neurodevelopmental conditions (e.g., history of Bell's palsy, history of four or more migraine headaches in the past 12 months that interfered with normal daily activity or any migraine headache in the past 5 years that required emergency or inpatient medical care, epilepsy, seizures in the last 5 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease). Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding treated basal cell and squamous cell carcinoma of the skin, which are allowed. Any autoimmune disease, including hypothyroidism without a defined non-autoimmune cause.
8. Any significant nasal or upper airway disease*.

   *(Including, but not limited to, being prone to epistaxis, a history of inflammatory rhinitis (including allergic rhinitis) that requires daily medications, cochlear implants, head/neck radiation history, anosmia/dysosmia, conditions that require prescription or over the counter intranasal medication (intermittent use will be allowed if no use occurred for 30 days before study vaccination and participant agrees to not use intranasal medication (other than steroids) for 30 days after study vaccination and to not use intranasal steroids for 6 months after study vaccination), and certain ear, nose and throat (ENT) conditions, including significant upper airway/nasopharyngeal disease or abnormal anatomy such as CSF leak.
9. Has an acute illness, as determined by the site PI or appropriate sub-investigator within 72 hours prior to study vaccination*.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
10. Has a positive test result for hepatitis B surface antigen, hepatitis C virus RNA (by reflex testing), or human immunodeficiency virus (HIV) antigen/antibody test at screening.
11. Has any confirmed or suspected immunosuppressive or immunodeficient state such as asplenia, recurrent severe infections and chronic* immunosuppressant medication within the past 6 months**.

    *Chronic meaning more than 14 continuous days.

    **Ophthalmic and topical steroids are allowed, see exclusion 19 for intranasal steroids.
12. Has received any investigational product within 60 days, or 5 half-lives, whichever is longer, before vaccination; or is planning to receive one during the study.
13. Has a history of hypersensitivity or severe allergic reaction* to any previous licensed or unlicensed vaccine or to the candidate vaccine components.

    * (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction)
    * See section 6.5.1 for vaccination formulation
14. Resides in or works in a nursing home or other skilled nursing facility.
15. Resides with or cares for immunocompromised persons, pregnant individuals, or children under 2 years of age (inclusive of health care workers and others with patient contact in health care settings).
16. People who handle rodents (laboratory workers, vivarium workers, pet store workers, etc.) or keep rodents as pets.
17. Received or plans to receive licensed inactivated/subunit vaccine within 14 days of study vaccine administration or live vaccine within 28 days of study vaccine administration.
18. Plan to receive a COVID-19 booster vaccine within the 180 days following study vaccination.
19. Regular use of intranasal medications including steroids*.

    *Participant must have had no intranasal medication use for 30 days prior to study vaccination and plans not to use intranasal medications for 30 days after study vaccination for medications other than steroids, and for 6 months after study vaccination for intranasal steroids (including over-the-counter Flonase).
20. Use of intranasal illicit drugs in the 5 years prior to study vaccination or plans to use during the study.
21. Planned international travel between vaccination and Day 29 visit.
22. Current smoker (including cigarettes, marijuana, and vaping) or smoking within 3 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Frequency of abnormal clinical safety laboratory AEs | Day 8
Frequency of solicited local adverse events (AEs) | Through Day 14 following vaccination
Frequency of systemic adverse events (AEs) | Through Day 14 following vaccination
Frequency of unsolicited AEs | Through Day 28 following vaccination
Occurrence of adverse events of special interest (AESIs) | Through Month 12 after vaccination
Occurrence of medically-attended adverse events (MAAEs) | Through Month 12 after vaccination
Occurrence of new-onset chronic medical conditions (NOCMCs) | Through Month 12 after vaccination
Occurrence of serious adverse events (SAEs) | Through Month 12 after vaccination
Severity of abnormal clinical safety laboratory AEs | Day 8
Severity of solicited local adverse events (AEs) | Through Day 14 following vaccination
Severity of systemic adverse events (AEs) | Through Day 14 following vaccination
Severity of unsolicited AEs | Through Day 28 following vaccination

SECONDARY OUTCOMES:
Geometric Mean Fold Rise (GMFR) of anti-vector antibodies | Through Day 366
Geometric Mean Fold Rise (GMFR) of mucosal anti-S binding antibodies (IgA, IgG) | Through Day 366
Geometric Mean Fold Rise (GMFR) of serum anti-S binding antibody (IgA and IgG) | Through Day 366
Geometric Mean Fold Rise (GMFR) of serum neutralizing antibodies to Spike variants | Through Day 366
Geometric Mean Titer (GMT) of anti-vector antibodies | Through Day 366
Geometric Mean Titer (GMT) of mucosal anti-S binding antibodies (IgA, IgG) | Through Day 366
Geometric Mean Titer (GMT) of serum anti-S binding antibody (Immunoglobulin A (IgA) and Immunoglobulin G (IgG )) | Through Day 366
Geometric Mean Titer (GMT) of serum neutralizing antibodies to Spike variants | Through Day 366
Median nasal swab quantitative polymerase chain reaction (qPCR) copy number for murine pneumonia virus (MPV) | Through Day 29
Percentage of participants positive for anti-vector antibodies | Through Day 366
Percentage of participants who seroconverted | Day 29
  Defined as a fourfold rise in serum neutralizing antibody titers
Percentage of participants with polymerase chain reaction (PCR)-positive nasal swab for murine pneumonia virus (MPV) | Through Day 29

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - NYU Grossman Long Island School of Medicine - Vaccine Center, Mineola, New York
  - Baylor College of Medicine, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT06441968/ICF_000.pdf